CLINICAL TRIAL: NCT04333186
Title: Expiratory Muscle Function in Critically Ill Ventilated Patients
Acronym: EMFIC
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Prof.dr. L.M.A. Heunks, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: EMFIC
Record Dates: First submitted 2020-03-29; First posted 2020-04-03 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Mechanical Ventilation; Expiratory Muscle; Critical Illness; Muscle Atrophy or Weakness; Diaphragm
MeSH Terms: conditions — Critical Illness; Muscular Atrophy; Asthenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data from ultrasound measurements — Data from ultrasound measurements and from the electronic patient record will be obtained / analyzed. One additional blood sample will be obtained within 24 hours after inclusion, during planned blood collection (from arterial line or venous puncture).

SUMMARY:
Inspiratory muscle weakness develops rapidly in ventilated critically ill patients and is associated with adverse outcome, including prolonged duration of mechanical ventilation and mortality. Surprisingly, the effects of critical illness on expiratory muscle function have not been studied.

The main expiratory muscles are the abdominal wall muscles, including the external oblique (EO), internal oblique (IO) and transversus abdominis muscles (TRA). These muscles are activated when respiratory drive or load increases, which can be during e.g. exercise, diaphragm fatigue, increased airway resistance, or positive airway pressure ventilation. The abdominal wall muscles are also critical for protective reflexes, such as coughing. Reduced abdominal muscles strength may lead to decreased cough function and thus inadequate airway clearance. This will lead to secretion pooling in the lower airways, atelectasis, and ventilator associated pneumonia (VAP). Studies have shown that decreased cough function is a risk for weaning failure and (re)hospitalization for respiratory complications. Further, high mortality was found in patients with low peak expiratory flow.

Considering the importance of a proper expiratory muscle function in critically ill patients, it is surprising that the prevalence, causes, and functional impact of changes in expiratory abdominal muscles thickness during mechanical ventilation (MV) for critically ill patients are still unknown.

Ultrasound is increasingly used in the ICU for the visualization of respiratory muscles. In a recent pilot study the investigators confirmed the feasibility and reliability of using of ultrasound to evaluate both diaphragm and expiratory abdominal muscle thickness in ventilated critically ill patients (manuscript in preparation). Accordingly, the primary aim of the present study is to evaluate the evolution of abdominal expiratory muscle thickness during MV in adult critically ill patients, using ultrasound data.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Invasive mechanical ventilation < 48 hours
* Expected duration of mechanical ventilation > 72 hours

Exclusion Criteria:

* Past medical history of neuromuscular disorders
* Mechanical ventilation > 48 hours within the current hospital admission
* Pregnant women
* Open abdominal wounds at proposed location of the ultrasound probe, due to recent abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient on mechanical ventilation in the intensive care
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Abdominal expiratory muscle thickness | From the date of inclusion until the date of first extubation or date of death from any cause, whichever came first, assessed up to 6 weeks
  Thickness of the abdominal expiratory muscles measured in millimeters

SECONDARY OUTCOMES:
Diaphragm muscle thickness | From the date of inclusion until the date of first extubation or date of death from any cause, whichever came first, assessed up to 6 weeks
  Thickness of the diaphragm muscle measured in millimeters
Inflammatory markers | Within 24 hours after inclusion
  Inflammatory markers (TNF-alpha, IL-6, IL-10) at inclusion (measured from blood sample using ELISA technique).
Applied driving pressure | From the date of inclusion until the date of first extubation or date of death from any cause, whichever came first, assessed up to 6 weeks
  Appplied driving pressuye defined as peak pressure minus total postive end expiratory pressure, and measured in centimetre of water
Tidal volume | From the date of inclusion until the date of first extubation or date of death from any cause, whichever came first, assessed up to 6 weeks
  Tidal volume measured in liters
Positive end expiratory pressure | From the date of inclusion until the date of first extubation or date of death from any cause, whichever came first, assessed up to 6 weeks
  Postive end expiratory pressure measure in centimetre of water
Extubation failure | From the date of extubation to the date of reintubation, or the date of death from any cause, or the date of ICU discharge, whichever came first, assessed up to 6 weeks
  Reintubated after extubation
Readmission to ICU | From the date of ICU diascharge to the date of death from any cause, or the date of hospital discharge, whichever came first, assessed up to 6 weeks
  Readmitted to ICU after the ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Leo M Heunks, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT04333186/Prot_SAP_000.pdf